CLINICAL TRIAL: NCT02658630
Title: Neurophysiological and Kinematic Predictors of Response in Chronic Stroke
Acronym: SRT4
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: VA Maryland Health Care System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N1667-R; HP-00062868 (Other: VA Maryland Healthcare Organization)
Record Dates: First submitted 2015-12-23; First posted 2016-01-20 (Estimated); Results first posted 2021-02-03 (Actual); Last update posted 2021-03-02 (Actual); Status verified 2021-02

CONDITIONS: Stroke
Keywords: arm rehabilitation; recovery of function
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Masking Description: The outcomes assessor is masked as to the prediction model and to particulars of performance during the intervention, but knows that there is a single group design.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Device: Robot + TTT Exercise (Experimental): All participants will be enrolled in this group to receive the same 60 minute study intervention consisting of wrist and shoulder-elbow robot training and TTT arm exercises.
  Interventions: Device: Robot + TTT exercise

INTERVENTIONS:
Device: Robot + TTT exercise — The intervention will be completed 36 visits approximately 3x/week for 12-18 weeks. The training progression will be sequential with 12 visits completed on the wrist robot, followed by 12 visits on the shoulder-elbow robot and completing with 12 visits alternating sessions on the wrist and shoulder-elbow robot. Participants will perform robot training for 45 minutes with each robot followed by 15 minutes of TTT practice to complete their 60 minute intervention session.

SUMMARY:
The purpose of this study is to design a predictive model of stroke recovery based on baseline measurements of arm movement and brain physiology. The expectation is the development of a formula to predict a person's response to an arm rehabilitation program provided in the chronic phase (6 months or greater post stroke) of recovery. The study will include magnetic resonance imaging (MRI), transcranial magnetic stimulation (TMS), genetic testing using blood and saliva, and an arm exercise program consisting of robot-assisted exercise combined with functional arm exercise called transition to task training (TTT).

DETAILED DESCRIPTION:
After informed consent, a baseline neurological exam, medical records review, MRI of the brain, TMS, questionnaires, cognitive testing, robot evaluations, and arm function testing will occur. Baseline testing will occur in the first 4-6 weeks of participation including two separate sessions approximately 1 week a part to examine arm strength, range of motion, and ability to perform functional tasks, with one additional session if needed to verify stability between results. Additionally, one robot evaluation, one MRI, and one TMS session will be completed. We will also collect genetic data using blood and saliva samples to examine potential RNA expression and genetic polymorphisms that might influence response to therapy.

The intervention phase consists of 12 weeks of robot and transition to task arm exercise training (TTT). Interventions will occur approximately 3 times per week for 12 weeks for a total of 36 visits. Additional time and visits will be allowed with visits occurring 4 times per week or up to 6 additional weeks (not to exceed 18 weeks) if scheduling conflicts arise. The intervention sessions will be one hour in duration.

During the hour-long intervention, 45 minutes of robotic intervention will be followed by 15 minutes of TTT. Two separate robots targeting different movements will be used for the 3 phases of the robot training. The training will be sequential with 12 sessions completed on the wrist robot, followed by 12 sessions on the shoulder-elbow robot and the final 12 sessions alternating between the wrist and elbow-shoulder robot.

After the final training session, subjects will return after a 12 week retention period. At various time points during and after the intervention phase there will be additional arm function testing, robot evaluations, questionnaires, blood draws, and TMS sessions to re-assess ability.

ELIGIBILITY:
Inclusion Criteria:

* Clinically defined, unilateral, hemiparetic stroke with radiologic exclusion of other possible diagnosis
* Stroke onset at least 6 months before enrollment
* Present with Mild/Moderate to Severe arm dysfunction (based on Fugl-Meyer scores of 10 to 45)
* Be medically stable to participate in the study and not have contractures or other impairments that would interfere with the interventional training.

Exclusion Criteria:

* Unable to give informed consent
* Have a serious complicating medical illness that would preclude participation.
* Contractures or orthopedic problems limiting range of joint motion in the potential study arm
* Visual loss such that the subject would not be able to see the test patterns on the robot computer monitor
* Botulinum toxin to study arm within four months of study enrollment or if received during the study period
* Unable to comply with requirements of the study
* Participants with a history of a seizure will not be precluded from the study, but will not be enrolled in the TMS portions
* Participants with electromagnetic exclusions (metal implants in the cranium, implanted electronic devices etc.) will not be precluded from the study but will be excluded from the MRI and TMS portions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2019-10-28 (Actual); Study Completion 2019-10-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George F. Wittenberg, MD PhD, Principal Investigator — VA Pittsburgh Healthcare System University Drive Division, Pittsburgh, PA
Locations (2):
- United States (2):
  - Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD, Baltimore, Maryland
  - VA Pittsburgh Healthcare System University Drive Division, Pittsburgh, PA, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
A de-identified, anonymized dataset will be created and shared. Where practicable, sharing should take place under a written agreement prohibiting the recipient from identifying or re-identifying (or taking steps to identify or re-identify) any individual whose data are included in the dataset. However, it is permissible for final datasets in machine-readable format to be submitted to and accessed from PubMed Central (and similar sites) provided that care is taken to ensure that the individuals cannot be re-identified using other publicly available information.
  Datasets will be made available to the public following appropriate approvals for disclosure criteria.
  Every effort will be made to protect personal privacy and the confidentiality of private information collected for research purposes. This particular dataset will be de-identified and the minimum amount of information necessary to achieve the objectives of the research proposed will be collected and shared.
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Derived] Dimyan MA, Harcum S, Ermer E, Boos AF, Conroy SS, Liu F, Horn LB, Xu H, Zhan M, Chen H, Whitall J, Wittenberg GF. Baseline Predictors of Response to Repetitive Task Practice in Chronic Stroke. Neurorehabil Neural Repair. 2022 Jul;36(7):426-436. doi: 10.1177/15459683221095171. Epub 2022 May 26. PMID 35616437

RESULTS

PARTICIPANT FLOW:
Recruitment Details: There were 68 participants consented. Of these 46 were eligible and entered the intervention. Four did not complete due to transportation issues, scheduling conflicts or lack of communication.
Period: Overall Study
Arm/Group | Device: Robot + TTT Exercise
Started | 46
Completed | 42
Not Completed | 4
Not completed — Withdrawal by Subject | 4

BASELINE CHARACTERISTICS:
Arm/Group | Device: Robot + TTT Exercise
Number analyzed (Participants) | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 27
  >=65 years | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.80952381 (11.2818397)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 42
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 23
  White | 19
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 42

OUTCOME MEASURES:

1. Primary Outcome: Stroke Impact Scale: Hand
Description: The Stroke Impact Scale (SIS) is one of the primary outcome measures assessing change in hand use from baseline testing to mid-training after visits 12 and 24, and post-training after visit 36 and the 12 week retention period. It is a self-report structured interview consisting of eight domains designed to assess physical, mental and emotional changes following stroke that contribute to quality of life. It has been tested and found to be reliable, valid, and sensitive to change in the stroke population. It has four physical domain subscales that can be analyzed separately. The SIS hand subscale will be the focus for our outcome measure. Higher scores indicate greater function and life satisfaction. The minimum and maximum for the subscale is 0 and 100 respectively.
Time Frame: Baseline, after visit 36, and 12 week retention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Device: Robot + TTT Exercise
Number analyzed (Participants) | 42
score on a scale
  Baseline | 20.4 (27.13)
  After visit 36 | 22.2 (24.26)
  12-week retention visit | 30.0 (30.57)

2. Primary Outcome: Fugl-Meyer Upper Extremity Assessment
Description: The Fugl-Meyer is one of the primary outcome measures assessing change in arm use from baseline testing to mid-training after visits 12 and 24, and post-training after visit 36 and the 12 week retention period. It is a stroke-specific measure of impairment of the upper extremity that has been shown to be valid and reliable with high inter-rater and test-retest reliability. It provides a direct-observational assessment of volitional movement and motor impairment related to reflexes, sensation, and abnormal synergies. Each item on the FM is rated on a three-point ordinal scale (0 = cannot perform, 1 = performs partially, 2 = performs fully). The scale ranges from 0-66 with higher scores representing less motor impairment.
Time Frame: Baseline, after visits 12, 24, and 36, and 12 week retention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Device: Robot + TTT Exercise
Number analyzed (Participants) | 42
score on a scale
  Baseline | 19.8 (9.62)
  After visit 12 | 22.2 (11.23)
  After visit 24 | 24.0 (13.08)
  After visit 36 | 24.4 (13.15)
  12-week retention | 25.2 (13.36)

3. Secondary Outcome: Action Research Arm Test (ARAT)
Description: The ARAT will be used to assess change from baseline testing to mid-training after visits 12 and 24, and post-training after visit 36 and the 12 week retention period. It is a stroke-specific measure of arm motor function and impairment of the upper extremity that has been shown to be valid and reliable with high inter-rater and test-retest reliability. It provides a direct-observational assessment of volitional movement. It includes 19 test activities and each test is given an ordinal score of 0, 1, 2, or 3, with higher values indicating better arm motor status. The total ARAT score is the sum of the 19 tests, and thus the maximum score is 57.
Time Frame: Baseline, after visits 12, 24, and 36, and 12 week retention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Device: Robot + TTT Exercise
Number analyzed (Participants) | 42
score on a scale
  Baseline | 14.4 (14.67)
  After visit 12 | 14.9 (15.33)
  After visit 24 | 16.2 (16.82)
  After visit 36 | 16.4 (16.57)
  12-week retention | 16.8 (17.73)

4. Secondary Outcome: 6-Item Wolf Motor Function Test (WMFT)
Description: The Streamlined 6-Item Wolf Motor Function Test (WMFT) will be used to assess change from baseline testing to mid-training after visits 12 and 24, and post-training after visit 36 and the 12 week retention period. It examines UE function based on task performance time, and quality of movement. Functional use and speed of movement are based on six timed activities. It has been examined in chronic stroke and has high inter-rater reliability, internal consistency, and test-retest reliability. Timed tasks that cannot be completed default to a time score of 120 seconds. Faster times or a lower score in seconds represent better function. The maximum score of 75 (minimum score 0) refers to perfect score on the full 15 item functional ability assessment (15 x 5.)
Time Frame: Baseline, after visits 12, 24, and 36, and 12 week retention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Device: Robot + TTT Exercise
Number analyzed (Participants) | 42
units on a scale
  Baseline | 1.7 (0.89)
  After visit 12 | 1.8 (1.08)
  After visit 24 | 1.9 (1.00)
  After visit 36 | 2.0 (1.13)
  12-week retention | 2.0 (1.20)

5. Other Pre Specified Outcome: TMS Score: Three Muscle Responses to Transcranial Magnetic Stimulation of the Motor Cortex
Description: TMS stimulation of the motor cortex will be performed using MagStim 200 Magnetic Stimulators (MagStim Ltd., Wales, UK) at baseline and post training after visit 36 and the 12 week retention to assess change in the motor evoked potential (MEP) of the arm muscles. TMS testing is as follows: 1) Location of muscle hotspot (highest motor evoked potential), 2) Threshold (lowest stimulation strength that evokes an MEP at hotspot) 3) Ipsilateral silent period measured on both the affected and unaffected side. A score on the scale of 0-9, 9 indicating a greater nervous system response.
Time Frame: Baseline, after visit 36, and 12 week retention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Device: Robot + TTT Exercise
Number analyzed (Participants) | 35
score on a scale
  Baseline | 2.4 (2.80)
  After visit 36 | 2.6 (3.03)
  12-week retention | 2.5 (3.09)

ADVERSE EVENTS:
Time Frame: 36 weeks
Arm/Group | Device: Robot + TTT Exercise
All-Cause Mortality (participants affected / at risk) | 0/42
Serious Adverse Events (participants affected / at risk) | 0/42
Other Adverse Events (participants affected / at risk) | 0/42

LIMITATIONS AND CAVEATS:
Total enrollment fell short of goals. There was some missing data in baseline measures, such as MRI or TMS.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-12): https://cdn.clinicaltrials.gov/large-docs/30/NCT02658630/Prot_SAP_000.pdf